CLINICAL TRIAL: NCT06545552
Title: Clinical Evaluation of the Efficacy and Safety of a Dietary Supplement on Hair Growth and Hair Health in Female With Acute Telogen Effluvium : a Double-blind, Randomized, Placebo-controlled, Clinical Study
Brief Title: Efficacy and Safety of a Dietary Supplement on Hair Growth and Hair Health in Female With Acute Telogen Effluvium
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Activ'inside (Industry)
Collaborators: Complife Italia Srl (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IT0000642/24 rev. 01
Record Dates: First submitted 2024-07-30; First posted 2024-08-09 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-06

CONDITIONS: Telogen Effluvium; Healthy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active product (Active Comparator): Hard shell capsule containing 280 mg of active compound.
  Interventions: Dietary Supplement: An oral formulation of green tea extract, bamboo shoot extract and selenium-enriched yeast
- Placebo (Placebo Comparator): Hard shell capsule containing maltodextrine
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: An oral formulation of green tea extract, bamboo shoot extract and selenium-enriched yeast — Hard shell capsule containing 280mg of the oral formulation
  Arms: Active product
Dietary Supplement: Placebo — Hard shell capsule containing maltodextrine
  Arms: Placebo

SUMMARY:
The study is aimed to assess the efficacy of a food supplement in reducing hair loss and accelerating the physiological growth in terms of elongation in female subjects showing acute telogen effluvium. Moreover, the efficacy of the product in increasing hair elasticity, thickness and brightness will be assess.

In order to reach this goal a randomized, double-blind, placebo controlled, parallel group (2 arms), clinical trial is carried out on 66 healthy female subjects aged between 18 and 52 years old, showing acute telogen effluvium will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Good general health
* Caucasian ethnicity
* All hair type included
* Transient acute telogen effluvium (duration less than 6 months) due to fatigue, seasonal change, deficiency of vitamins and minerals, stress, change or imbalance of normal daily routing, or emotional stress
* Subjects having a positive pull test result
* Subjects with minimum hair length of 6/7 cm
* Subjects who stopped any anti hair loss treatment at least 3 months prior the study
* Subjects agreeing not to take any treatment (oral or topic) able to interfere with the hair growth, diameter or fall during the whole study duration
* Willingness not to dye/blench hair during the 2 weeks preceding each visit
* Willingness not to cut hair for all the study length
* Subjects registered with health social security or health social insurance
* Subjects having signed their written Informed Consent form (ICF) and Privacy Policy for their participation in the study and a photograph authorization
* Subjects able to understand the language used in the investigation centre and the information given
* Subjects able to comply with the protocol and follow protocol constraints and specific requirements
* Willingness to use during all the study period only the product to be tested
* Willingness not to use similar products that could interfere with the product to be tested
* Willingness to not vary the normal daily routine (i.e. lifestyle, physical activity, diet etc.)
* Subjects under effective contraception (oral/not oral) if women of childbearing potential; not expected to be changed during the trial

Exclusion Criteria:

* Subjects who do not meet the inclusion criteria
* Subject is taking part or planning to participate to another clinical study in the same or in another investigation centre
* Subject who is deprived of freedom by administrative or legal decision or under guardianship
* Subject admitted in a sanitary or social facilities
* Subject who is planning a hospitalization during the study
* Subjects under treatment with food supplements which could interfere with the functionality of the product under study
* Subject has participated in another clinical study with anti-hair loss product or treatment within the last 24 weeks before the inclusion visit
* Subject breastfeeding, pregnant or not willing to take necessary precautions to avoid pregnancy during the study (if women of childbearing potential)
* Subject has started or changed oestrogen-progesterone contraception or hormonal treatment, within the 3 months prior to the study or foreseeing it for the duration of the study
* Subject having an acute, chronic or progressive illness liable to interfere with the study data or considered by the Investigator hazardous for the subject or incompatible with the study requirements
* Subjects under radiotherapy, chemotherapy at any time
* Subjects under locally pharmacological/non-pharmacological treatment applied on the area of interest monitored during the test
* Subject having food disorders
* Subject who has any other hair disorder or hair disease (female pattern hair loss, any type of alopecia…)
* Subject having excessive and/or fluctuating hair shedding for more than 6 months
* History or clinical signs of hyperandrogenaemia
* Systemic treatment affecting the hair growth taken for more than 4 consecutive weeks during the last 24 weeks before inclusion visit
* Systemic or local androgenetic alopecia treatment or product, taken or applied (Minoxidil, Aminexil, Finasteride, Dutasteride, cosmetic solution or capsules with vitamin B, zinc, caffeine…) for more than 4 consecutive weeks during the last 24 weeks before the inclusion visit
* Any hair care product applied on the scalp between the last shampoo and the inclusion visit (e.g. gel, hairspray, wax, foam…)
* Scalp surgery (hair transplants, laser) at any time.
* Not menopausal women

Ages: 18 Years to 52 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 66 (Actual)
Dates: Start 2024-09-30 (Actual); Primary Completion 2025-01-24 (Actual); Study Completion 2025-01-24 (Actual)

PRIMARY OUTCOMES:
Change in Anagen hair density | after 84 days of supplementation
  Number of hairs in anagen phase per cm² and proportion (in %) using phototricogram (TrichoScan)

SECONDARY OUTCOMES:
Change in hair brightness | after 42 and 84 days of supplementation
  8° gloss value (average value of 5 measures) using spectrophotometer/colorimeter CM 700D (Konica-Minolta).
Change in hair elasticity | after 42 and 84 days of supplementation
  using a dynamometer (Tensolab 2512A, Mesdan Lab)
Change in hair volume | after 42 and 84 days of supplementation
  Using a 7-point scale administred by a dermatologist
Change in hair loss | after 42 and 84 days of supplementation
  Number of extracted hairs using a pull test
Change in Total Hair Density | after 42 and 84 days of supplementation
  Number of total hairs per cm² using phototricogram (TrichoScan)
Change in Telogene Hair Density | after 42 and 84 days of supplementation
  Number of hairs in telogen phase per cm² and proportion (in %) using phototricogram (TrichoScan)
Change in Anagen hair density | after 42 days of supplementation
  Number of hairs in anagen phase per cm² and proportion (in %) using phototricogram (TrichoScan)

CONTACTS AND LOCATIONS:
Overall Officials: Gloria Roveda, MD, PhD, Principal Investigator — Complife Italia srl Via Mons. Angelini, 21 27028 San Martino Siccomario (PV)
Locations (1):
- Complife Italia srl, San Martino Siccomario, Italy

IPD SHARING:
Plan to Share IPD: No